CLINICAL TRIAL: NCT02062281
Title: A Phase 4, Randomized, Single-blind Trial to Evaluate Safety and Immunogenicity of a 23-Valent Pneumococcal Polysaccharide Vaccine When Administered Simultaneously With Trivalent Inactivated Influenza Vaccine in Healthy Children Aged 3-7years and Healthy Adults 65 Aged 50-65years.
Brief Title: Study of Evaluating Safety and Immunogenicity of 23-Valent Pneumococcal Polysaccharide Vaccine With Influenza Vaccine in Children and Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Chengdu Institute of Biological Products Co.,Ltd. (Industry); Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JSEPI-002
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Pneumococcal Infection; Influenza
Keywords: Safety; Immunogenicity; vaccine; pneumococcal; influenza
MeSH Terms: conditions — Pneumococcal Infections; Influenza, Human | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 23-valent Pneumococcal Polysaccharide vaccine (Active Comparator): 0.5ml 23-valent pneumococcal Polysaccharide vaccine made by Chengdu Institute of Biological Products Co.,Ltd.
  lot number: 20130106-1, duration:JAN,17,2015.
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine
- Trivalent Influenza Vaccine (Active Comparator): 0.5ml trivalent influenza vaccine made by Shanghai Institute of Biological Products Co.,Ltd.
  lot number:20130713, duration:Jul,1,2014.
  Interventions: Biological: trivalent influenza vaccine
- 23vPPV+TIV (Experimental)
  Interventions: Biological: 23vPPV+TIV

INTERVENTIONS:
Biological: 23-valent pneumococcal polysaccharide vaccine — Single 0.5ml 23-valent pneumococcal polysaccharide vaccine was administered intramuscularly (IM)
  Arms: 23-valent Pneumococcal Polysaccharide vaccine
Biological: trivalent influenza vaccine — Single 0.5ml trivalent influenza vaccine was administered IM
  Arms: Trivalent Influenza Vaccine
Biological: 23vPPV+TIV — Single 0.5 ml 23-valent pneumococcal polysaccharide vaccine (23vPPV) and a single 0.5 ml trivalent inactivated influenza vaccine (TIV) were administered IM, in one day.
  Arms: 23vPPV+TIV

SUMMARY:
The 23-valent pneumococcal Polysaccharide vaccine (23vPPV) has been developed for children and adults to prevent pneumococcal diseases such as pneumonia (inflammation of the lungs), meningitis (inflammation of the brain lining), and septicemia (blood poisoning) since 2006 in China. Also, the trivalent influenza vaccine (TIV) is frequently administered to the children and adults. The main objective of this study is to show that both vaccines can safely be administered together without affecting the immune response of protecting against disease.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy male or female, for adults 50-65 years of age, for children 3-7 years of age.
2. Available for the duration of the trial - approximately 2 months.
3. No history of severe adverse reaction associated with a vaccine.

Exclusion Criteria:

1. Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc.
2. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain.
3. Autoimmune disease or immunodeficiency.
4. Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids.
5. Diabetes mellitus (type I or II), with the exception of gestational diabetes History of thyroidectomy or thyroid disease that required medication within the past 12 months.
6. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.
7. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
8. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
9. History of any blood products or seasonal influenza vaccine administration within 3 months before the dosing.
10. Administration of any other investigational research agents within 30 days before the dosing.
11. Administration of any live attenuated vaccine within 30 days before the dosing Administration of subunit or inactivated vaccines, e.g., pneumococcal vaccine, or allergy treatment with antigen injections, within 14 days before the dosing.
12. Axillary temperature > 37.0 centigrade at the time of dosing.
13. Psychiatric condition that precludes compliance with the protocol.
14. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2225 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of 23vPPV | 1 month after 23vPPV vaccination
  IgG GMC measured by enzyme-linked immunosorbent assay (ELISA) and expressed in micrograms per mL (mcg/mL) for serotypes 1,2,5,6B,14,19F,23F,which were frequently detected in patients in Chinese.
Immunogenicity of TIV | 1 month after TIV vaccination
  Percentage of participants achieving at Least a 4-fold Increase in the Titer of the Standard Hemagglutination Inhibition Assay (HAI)

SECONDARY OUTCOMES:
adverse events following the immunization (AEFI) | 28 days after 23vPPV and TIV vaccination

CONTACTS AND LOCATIONS:
Overall Officials: ma fubao, doctor, Principal Investigator — Jiangsu CDC
Locations (1):
- Yangzhong Center for Disease Control and Prevention, Zhenjiang, Jiangsu, China